CLINICAL TRIAL: NCT06254651
Title: Resuscitation Table Height for Face-mask Ventilation in Infants
Acronym: ForTab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEOUNIPD4(2023)
Record Dates: First submitted 2023-12-01; First posted 2024-02-12 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Asphyxia; Resuscitation; Newborn Morbidity
MeSH Terms: conditions — Asphyxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High resuscitation table (Experimental): Participants will be invited to administer face-mask ventilation setting the table height to the operator's xiphoid process in a neonatal manikin.
  Interventions: Other: High resuscitation table
- Low resuscitation table (Active Comparator): Participants will be invited to administer face-mask ventilation setting the table height to the operator's superior anterior iliac spines in a neonatal manikin.
  Interventions: Other: Low resuscitation table

INTERVENTIONS:
Other: High resuscitation table — Participants will be invited to administer face-mask ventilation setting the table height to the operator's xiphoid process in a neonatal manikin.
  Arms: High resuscitation table
Other: Low resuscitation table — Participants will be invited to administer face-mask ventilation setting the table height to the operator's superior anterior iliac spines in a neonatal manikin.
  Arms: Low resuscitation table

SUMMARY:
Positive pressure ventilation (PPV) is the most important intervention in neonatal resuscitation. During PPV, it is important to hold the face-mask with care, as applying excessive pressure could cause injury to the infant, while insufficient pressure could be a contributor of mask leak and reduced effective ventilation. Application of positive pressure to face structures may trigger a vagally mediated reflex via the trigeminal nerve that innervates the skin of the face leading to apnoea and a decrease in heart rate (TCR, trigeminal-cardiac reflex).

The force exerted by providers during neonatal ventilation to improve mask seal might result in pressure lesions and the elicitation of the trigeminal-cardiac reflex. The height of the resuscitation could influence the forces applied to the face and the quality of the procedure. Information about the applied forces in relation to the height of the resuscitation table is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Level III neonatal intensive neonatal care unit consultants and pediatric residents

Exclusion Criteria:

* None

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Applied forces on the manikin face | 1 minute after initiation of ventilation
  The forces applied by the participants to the manikin face will be measured by sensors positioned on the manikin face

SECONDARY OUTCOMES:
Cuff pressure | 1 minute after initiation of ventilation
  The pressure inside the mask will be measured during the procedure
Percentage of ventilation time with leak less than 25% around the mask | 1 minute after initiation of ventilation
  The mask leak will be measured by using a respiratory function monitoring during the procedure

OTHER OUTCOMES:
Participants' opinion on the procedures | 5 minutes after the end of the procedure
  Participants will be asked to rate both procedures by using a Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Padova, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madar J, Roehr CC, Ainsworth S, Ersdal H, Morley C, Rudiger M, Skare C, Szczapa T, Te Pas A, Trevisanuto D, Urlesberger B, Wilkinson D, Wyllie JP. European Resuscitation Council Guidelines 2021: Newborn resuscitation and support of transition of infants at birth. Resuscitation. 2021 Apr;161:291-326. doi: 10.1016/j.resuscitation.2021.02.014. Epub 2021 Mar 24. PMID 33773829
- [Background] Wyckoff MH, Wyllie J, Aziz K, de Almeida MF, Fabres JW, Fawke J, Guinsburg R, Hosono S, Isayama T, Kapadia VS, Kim HS, Liley HG, McKinlay CJD, Mildenhall L, Perlman JM, Rabi Y, Roehr CC, Schmolzer GM, Szyld E, Trevisanuto D, Velaphi S, Weiner GM; Neonatal Life Support Collaborators. Neonatal Life Support 2020 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Resuscitation. 2020 Nov;156:A156-A187. doi: 10.1016/j.resuscitation.2020.09.015. Epub 2020 Oct 21. PMID 33098917
- [Background] Schilleman K, Witlox RS, Lopriore E, Morley CJ, Walther FJ, te Pas AB. Leak and obstruction with mask ventilation during simulated neonatal resuscitation. Arch Dis Child Fetal Neonatal Ed. 2010 Nov;95(6):F398-402. doi: 10.1136/adc.2009.182162. Epub 2010 Jun 30. PMID 20591880
- [Background] van Vonderen JJ, Kleijn TA, Schilleman K, Walther FJ, Hooper SB, te Pas AB. Compressive force applied to a manikin's head during mask ventilation. Arch Dis Child Fetal Neonatal Ed. 2012 Jul;97(4):F254-8. doi: 10.1136/archdischild-2011-300336. Epub 2011 Dec 5. PMID 22147285
- [Background] Cavallin F, Sala C, Maglio S, Bua B, Villani PE, Menciassi A, Tognarelli S, Trevisanuto D. Applied forces with direct versus indirect laryngoscopy in neonatal intubation: a randomized crossover mannequin study. Can J Anaesth. 2023 May;70(5):861-868. doi: 10.1007/s12630-023-02402-9. Epub 2023 Feb 14. PMID 36788198
- [Background] Lee HC, Yun MJ, Hwang JW, Na HS, Kim DH, Park JY. Higher operating tables provide better laryngeal views for tracheal intubation. Br J Anaesth. 2014 Apr;112(4):749-55. doi: 10.1093/bja/aet428. Epub 2013 Dec 18. PMID 24355831
- [Derived] Zamunaro A, Cavallin F, Maglio S, Villani PE, Bua B, Gallo D, Menciassi A, Tognarelli S, Trevisanuto D. Applied forces with high vs. low resuscitation table during neonatal ventilation: a randomized crossover manikin study. Eur J Pediatr. 2024 Nov 27;184(1):45. doi: 10.1007/s00431-024-05844-5. PMID 39592514